CLINICAL TRIAL: NCT04185649
Title: A Clinical Study Evaluating the Efficacy and Safety of BAT8001 Injection for the Treatment of HER2-positive Advanced Breast Cancer - A Multicenter, Randomized, Open-label, Positive-controlled, Superiority Phase III Clinical Trial in China
Brief Title: The Efficacy and Safety of BAT8001 Injection for the Treatment of HER2-positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8001-002-CR
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HER2-positive Advanced Breast Cancer
MeSH Terms: interventions — Injections; Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT8001 for injection (Experimental): Participants with HER2-positive, unresectable LABC or MBC who have experienced disease progression after treatment with trastuzumab and a taxane will be treated with trastuzumab emtansine. Participants may continue to receive study treatment until disease progression (as assessed by the investigator), unmanageable toxicity, or study termination by the Sponsor.
  Interventions: Biological: BAT8001 for injection
- Control (lapatinib + capecitabine) (Active Comparator): Participants with HER2-positive, unresectable LABC or MBC who have experienced disease progression after treatment with trastuzumab and a taxane will be treated with lapatinib plus capecitabine. Participants may continue to receive study treatment until disease progression (as assessed by the investigator), unmanageable toxicity, or study termination by the Sponsor.
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Biological: BAT8001 for injection — 3.6 mg/kg, q3w, administered intravenously on day 1 of each treatment cycle, 21 days/treatment cycle.
  Arms: BAT8001 for injection
Drug: Lapatinib — Lapatinib 1250 mg was administered orally once per day of each 21-day cycle.
  Other Names: Lapatinib ditosylate tablets
  Arms: Control (lapatinib + capecitabine)
Drug: Capecitabine — Capecitabine 1000 milligrams per square meter (mg/m^2) was administered orally twice daily on Days 1-14 of each 21-day cycle.
  Other Names: capecitabine tablets
  Arms: Control (lapatinib + capecitabine)

SUMMARY:
To evaluate the safety and efficacy of BAT8001 for the treatment of HER2-positive advanced breast cancer, using lapatinib in combination with capecitabine as the positive control drug.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, positive-controlled, superiority phase III clinical study. The object is to evaluate the safety and efficacy of BAT8001 for the treatment of HER2-positive advanced breast cancer, using lapatinib in combination with capecitabine as the positive control drug.

Eligible subjects will be randomized to the experimental or control group in a 1:1 ratio and stratified by the number of HER2-positive advanced/metastatic breast cancer treatment regimens (0, 1 VS > 1) and lesion site (organ VS non-organ).

ELIGIBILITY:
Inclusion Criteria:

1. Patients are required to provide at least 10 unstained sections.
2. HER2-positive (defined as: IHC 3+ or FISH+) confirmed by the central laboratory of this study.
3. Histologically and/or cytologically confirmed invasive breast cancer, including unresectable locally advanced breast cancer (LABC) or metastatic breast cancer (MBC).
4. LABC or MBC that has progressed during or after treatment, or during or within 12 month following adjuvant therapy as confirmed by imaging.
5. Previously received adjuvant therapy, or locally advanced/metastatic breast cancer treatment regimen that included taxanes and trastuzumab (including approved biosimilars) as monotherapy or combination therapy。
6. At least one measurable lesion or a single metastatic tumor in the bone as per the Response Evaluation Criteria in Solid Tumor (RECIST) 1.1.
7. A score of 0-1 for performance status as per the Eastern Cooperative Oncology Group (ECOG) scale.
8. Expected survival ≥ 3 months.
9. Left ventricular ejection fraction (LVEF) ≥ 50%.
10. If anthracyclines are used, the cumulative dose must meet the following criteria: the cumulative dose must not exceed the equivalent dose of doxorubicin 500 mg/m2.
11. Women of childbearing age or fertile male subjects must agree to use oral, implanted, or injectable hormone contraceptives as well as one or two forms of non-hormonal contraceptive measures during the study period and until 6 months after the end of the study.
12. Blood pregnancy test must indicate non-pregnant for all women of childbearing potential and those who do not meet the definition of postmenopause.

Exclusion Criteria:

1. Current presence of grade ≥ 2 peripheral neuropathy.
2. History of other malignant tumors within the past 5 years, but does not include properly treated cervical carcinoma in situ, non-melanoma skin cancer, stage 1 uterine cancer, or other tumors with good prognosis.
3. Received treatment with a cancer drug or investigational drug within 21 days from the first dose of the study drug, except for hormone therapy..
4. Received radiation therapy within 14 days prior to the first test drug administration of this study; or subject has not recovered from the acute toxicity of radiation therapy prior to the first test drug administration of this study.
5. Brain metastasis that is symptomatic or requires treatment to control symptoms within 30 days before randomization.
6. Subjects who must receive the first test drug administration within less than 14 days following the completion of radiation therapy for symptomatic brain metastasis.
7. Currently experiences moderate or severe dyspnea at rest caused by advanced malignancy or other complications or severe primary lung diseases, or currently requires continuous oxygen therapy, or subject currently suffers from interstitial lung disease (ILD) or pneumonia/pneumonitis.
8. History of myocardial infarction or unstable angina within 6 months prior to first test drug administration.
9. Previous history of LVEF falling below 40%; or presence of symptomatic congestive heart failure (CHF) during trastuzumab (including other analogues) treatment.
10. Symptomatic congestive heart failure (CHF; New York Heart Association [NYHA] Class II-IV); Severe arrhythmias requiring treatment.
11. Presence of severe and uncontrollable systemic diseases (e.g. clinically significant cardiovascular, lung or metabolic diseases).
12. Patients who currently require coumarin derivative-based anticoagulation therapy such as warfarin and phenprocoumon.
13. Presence of diseases that may affect intestinal absorption, including malabsorption syndrome, stomach and small bowel resection, and ulcerative colitis.
14. Intolerance (grade 3-4 infusion reactions) or allergy to trastuzumab (and other analogues) or mouse proteins or any ingredient of the medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 18 months
  PFS is defined as the time from randomization to the first occurrence of disease progression as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) Version (v1.1), or death from any cause during the study, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 30 months
  OS is defined as the time from the date of randomization to the date of death from any cause.
Objective Response Rate (ORR) | Up to approximately 30 months
  ORR is defined as percentage of participants with partial response (PR) or complete response (CR) determined on the basis of investigator assessments with the use of RECIST v1.1.
Duration of Response (DOR) | Up to approximately 30 months
  DOR is defined as as the time from the date of initial confirmed PR or CR to the date of disease progression or death within the study.
Clinical Benefit Rate (CBR) | Up to approximately 30 months
  CBR is defined as the proportion of subjects with best overall response (confirmed PR or CR) or with stable disease (confirmed SD) for at least 6 months;
Serum Concentration of BAT8001 | Pre-dose and 15-30 minutes after dose on Day 1, Day 8, Day 15 of each 21-day cycle during Cycles 1-4 and at completion/early termination visit (up to approximately 30 months)
  Concentration of BAT8001 will be measured in serum from participants, who received BAT8001.
Serum Concentration of total antibody of BAT8001 for injection | Pre-dose and 15-30 minutes after dose on Day 1, Day 8, Day 15 of each 21-day cycle during Cycles 1-4 and at completion/early termination visit (up to approximately 30 months)
  Concentration of total antibody will be measured in serum from participants, who received BAT8001.
Plasma Concentration of batansine (a maytansine derivative, which is the 3AA-MDC complex) | Pre-dose and 15-30 minutes after dose on Day 1, Day 8, Day 15 of each 21-day cycle during Cycles 1-4 and at completion/early termination visit (up to approximately 30 months)
  Concentration of batansine will be measured in plasma from participants, who received BAT8001.
Percentage of Participants with Anti-therapeutic Antibodies (ATA) to BAT8001 | Pre-dose on Day 1 of each 21-day cycle during Cycles 1-4 and at completion/early termination visit (up to approximately 30 months)
  ATA to BAT8001 were measured in serum of participants, who received BAT8001.

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, M.D., Principal Investigator — Sun Yat-sen University
Locations (51):
- China (51):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking union medical college hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Foshan City No. 1 People's Hospital, Foshan, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital. SYSU, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-sen University, Zhuhai, Guangdong
  - Liuzhou workers hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of science and technology, Luoyang, Henan
  - The First Affiliated Hospital of Xixiang Medical College, Xinxiang, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College of HUST, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Yichang Central Hospital, Yichang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanning, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Yancheng City No. 1 People's Hospital, Yancheng, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The Second Hospital of Anhui Medical University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hispotal of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No